CLINICAL TRIAL: NCT05349799
Title: A Prospective, Multicentric, Open-labelled, Interventional Study to Assess Skin Beautification by Treating Fine Lines in the Neck, Perioral and Smiling Lines Areas With TEOSYAL RHA® 1
Brief Title: TEOSYAL RHA® 1 for Neck Lines, Perioral Lines and Smiling Lines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEO-RHAR1-2005
Record Dates: First submitted 2022-04-20; First posted 2022-04-27 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Skin Aging; Fine Lines of the Face and Neck
MeSH Terms: interventions — Needles; Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEOSYAL RHA® 1 (Experimental): Subjects injected with TEOSYAL RHA® 1 during the "skin beautification" phase, not further treated with TEOSYAL® PureSense Redensity 1 during the "skin redensification" phase.
  Interventions: Device: TEOSYAL RHA® 1
- TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 with a needle (Experimental): Subjects injected with TEOSYAL RHA® 1 during the "skin beautification" phase, further treated with TEOSYAL® PureSense Redensity 1 using a needle during the "skin redensification" phase.
  Interventions: Device: TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 (needle)
- TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 with a cannula (Experimental): Subjects injected with TEOSYAL RHA® 1 during the "skin beautification" phase, further treated with TEOSYAL® PureSense Redensity 1 using a cannula (optional for perioral lines) during the "skin redensification" phase.
  Interventions: Device: TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 (cannula)

INTERVENTIONS:
Device: TEOSYAL RHA® 1 — During the first phase of the study, ubjects will be treated with TEOSYAL RHA® 1 at baseline (V1) and may receive an optional treatment at 1 month (V2).
  In the exploratory phase of the study, subjects will not receive any additional treatment.
  Arms: TEOSYAL RHA® 1
Device: TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 (needle) — During the first phase of the study, ubjects will be treated with TEOSYAL RHA® 1 at baseline (V1) and may receive an optional treatment at 1 month (V2).
  In the exploratory phase of the study, subjects will receive additional treatment with TEOSYAL® PureSense Redensity 1 using a needle. TEOSYAL® PureSense Redensity 1 will be administered over three sessions at 2, 3 and 4 months after baseline (respectively V3, V4 and V5).
  Arms: TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 with a needle
Device: TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 (cannula) — During the first phase of the study, ubjects will be treated with TEOSYAL RHA® 1 at baseline (V1) and may receive an optional treatment at 1 month (V2).
  In the exploratory phase of the study, subjects will receive additional treatment with TEOSYAL® PureSense Redensity 1 using a cannula. TEOSYAL® PureSense Redensity 1 will be administered over three sessions at 2, 3 and 4 months after baseline (respectively V3, V4 and V5).
  Arms: TEOSYAL RHA® 1 and TEOSYAL® PureSense Redensity 1 with a cannula

SUMMARY:
Prospective, low-interventional, multicentric, open-labelled study to assess the performance and safety of skin beautification treatment by TEOSYAL RHA® 1 for fine lines in the neck, perioral region, and smiling lines including an exploratory arm with TEOSYAL® PureSense Redensity 1 to assess skin redensification.

Treatment phase - skin beautification:

At Visit 1 (Baseline), subjects will be injected with TEOSYAL RHA® 1 in the fine lines (Neck lines and Perioral and/or Smiling lines) depending on wrinkle severity assessed by the Principal Investigator (PI) at baseline using a specific grading scale for each indication.

The subject will be included in the study if he has been graded 2 or 3 on the Neck Lines Descriptive Scale (NLDS) at baseline.

Then:

1. The subject will be included in the perioral rhytids cohort if he has been graded 2 or 3 on the Perioral Rhytids Severity Rating Scale (PR-SRS) at baseline.
2. The subject will be included in the smiling lines cohort if he has been graded 3 or 4 on the Smiling Lines Descriptive Scale (SLDS) at baseline.

Each indication represent one cohort and all subjects will be included in the neck lines cohort.

Thus, Subject participating to the study may be treated for:

* Neck Lines and perioral Lines (2 cohorts)
* Neck Lines and Smiling Lines (2 cohorts)
* Neck Lines, Perioral Lines and Smiling Lines (3 cohorts)

An optional touch-up will be performed at Visit 2 (Month 1 +/- 1 week) if deemed necessary to achieve an optimal correction.

Exploratory phase - skin redensification:

After treatment with TEOSYAL RHA® 1, subjects will be randomized to the second phase of the study (starting at month 2 +/- 1 week): 5/6 of the subjects will enter the exploratory part of the study during which TEOSYAL® PureSense Redensity 1 (RHA1+R1 treated Group) will be assessed for skin redensification. The rest of the subjects will not receive any additional treatment for the rest of the study (RHA1 only treated group/around 11 subjects).

Note: the number of sessions treated with Redensity 1 might be adapted depending on subject treatment needs in order to achieve optimal results. This will be at PI discretion.

Subjects in the RHA+R1 treated Group will be also randomized into 2 subgroups of 28 subjects as described below:

* Sub-Group A: injection with a needle for all indications
* Sub-Group B: injection with a cannula for neck lines and smiling lines indications* *The perioral indication will be treated with a needle for this group.

The principal investigator (PI) will perform the study injections. He will evaluate subject aesthetic improvement using grading scales and skin quality measurements at each study visits and assess safety and tolerability of the devices during the study. Adverse events will be monitored by the Clinical Research Associate (CRA) throughout the study.

Additionally, a Blinded Evaluator will also evaluate subject aesthetic improvement using grading scales for each follow-up visits based on photographs.

ELIGIBILITY:
Inclusion Criteria (General):

1. Healthy adults, 35 to 70 years old seeking an improvement of their aesthetic appearance and beautification of their skin in 3 areas: perioral lines, smiling lines and neck lines.
2. Subjects having given their informed consent.
3. Subjects having wrinkle severity ranked as mild to moderate neck lines (grade 2 or grade 3 on the NLDS)

Inclusion Criteria (Cohort) 4. Healthy adult having wrinkle severity in at least one of the two indications (50% for each of the following cohort): i. Moderate to severe perioral rhytids (grade 2 or grade 3 on the PR-SRS) ii. Moderate to severe smiling lines (grade 3 or grade 4 on the SLDS)

Exclusion Criteria:

1. Minor subjects
2. Subjects who already had fillers and/or other skin quality treatment(s) in the 6 months preceding the study.
3. Subjects undergoing or planning to undergo peeling treatment or laser/ultrasound-based treatment during the study or having had one of these treatments in the 6 months preceding the study.
4. Subjects showing cutaneous disorders, inflammation or infection (acne, herpes, scars…) at the treatment site or near to this site.
5. Subjects having a known hypersensibility to lidocaine and/or amide local anesthetic agents or hyaluronic acid, or with history of severe allergy or anaphylactic shock.
6. Subjects with autoimmune or cardiac diseases and/or undergoing treatment for heart diseases (beta blockers).
7. Subjects with hepatocellular insufficiency and/or undergoing treatment for liver disease.
8. Subjects suffering from epilepsy or porphyria.
9. Subjects with severe, ongoing and/or uncontrolled disease that may pose a health risk to the subject during the study and/or may have an impact on the study assessments.
10. Subjects receiving or planning to receive high dose Vitamin E, aspirin, anti-inflammatories, or anti-coagulant during the week preceding each injection.
11. Subjects receiving any long-term medical treatment or any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject at undue risk.
12. Subjects under guardianship/tutorship.
13. Pregnant women or breastfeeding mother.
14. Subjects participating to another research on human beings or being in an exclusion period for a previous study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects improved or much improved on the Global Aesthetic Improvement Scale (GAIS) according to both the Principal Investigator (PI) and the subject. | Visit 3 (Month 2)
  The Global Aesthetic Improvement Scale (GAIS) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".

SECONDARY OUTCOMES:
Proportion of subjects improved or much improved on the Global Aesthetic Improvement Scale (GAIS) according to the Principal Investigator (PI) | Visit 2 (Month 1), Visit 3 (Month 2), Visit (Month 3), Visit 5 (Month 4), Visit 6 (Month 5)
  The Global Aesthetic Improvement Scale (GAIS) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
Proportion of subjects improved or much improved on the Global Aesthetic Improvement Scale (GAIS) according to the subject | Visit 2 (Month 1), Visit 3 (Month 2), Visit (Month 3), Visit 5 (Month 4), Visit 6 (Month 5)
  The Global Aesthetic Improvement Scale (GAIS) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
Proportion of subjects improved or much improved on the Global Aesthetic Improvement Scale (GAIS) according to the Blinded Evaluator (BE) | Visit 2 (Month 1), Visit 3 (Month 2), Visit (Month 3), Visit 5 (Month 4), Visit 6 (Month 5)
  The Global Aesthetic Improvement Scale (GAIS) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Site 4, Alicante
  - Site 3, Barcelona
  - Site 1, Bilbao
  - Site 2, Madrid

IPD SHARING:
Plan to Share IPD: No